CLINICAL TRIAL: NCT07332039
Title: The Effect of Watching Cat Videos on Maternal Stress and Fetal Well-being: A Single-Blind Randomized Controlled Trial
Brief Title: The Effect of Watching Cat Videos on Non-Stress Test Results And Stress Parameters in Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Rukiye Duman, Research assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IstanbulUC-EBE-RD-02
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Maternal Stress; Fetal Well-Being
Keywords: Fetal Well-Being; Maternal Stress; Cat Videos

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Participants randomly assigned to the control group will also rest in a private room for 10 minutes, after which all initial measurements will be taken. A routine NST will then be performed.
  Interventions: Behavioral: Non-Video Watching Group
- Intervention group (Experimental)
  Interventions: Behavioral: Group watching cat videos

INTERVENTIONS:
Behavioral: Group watching cat videos — The cat video, which will be shown to pregnant women as part of the study, will be implemented as an intervention to reduce participants' stress levels during the NST. The NST session takes approximately 20 minutes, and the video will be played for this duration. The content of the video will be carefully selected to create a relaxing and entertaining effect on the audience. Participants will begin watching the video immediately after connecting to the NST device and will continue to watch throughout the NST. This process aims to calm participants, reduce stress levels, and promote overall relaxation.
  Arms: Intervention group
Behavioral: Non-Video Watching Group — Participants randomly assigned to the control group will also rest for 10 minutes in a private room and all initial measurements will be taken.
  Arms: Control Group

SUMMARY:
Pregnancy is a period in which women are physiologically and psychologically vulnerable, and the stress experienced can affect both maternal mental health and fetal well-being. The non-stress test (NST), used to assess fetal health in the final weeks of pregnancy, can cause anxiety in some women because it requires the mother to remain supine and immobile for extended periods. Prolonged testing or non-reactive results can also increase this stress. Therefore, simple methods are needed to reduce stress during NST. Humorous and cute content, especially animal videos, is known to promote positive emotions and psychological relaxation. This study evaluated the effects of watching cat videos during NST on stress levels and fetal physiological parameters in primiparous pregnant women.

DETAILED DESCRIPTION:
Pregnancy is a sensitive period during which women experience a variety of changes, both physiologically and psychologically. Stress factors encountered during this period can negatively impact the mother's mental health and fetal well-being. Non-stress testing (NST) is a non-invasive screening method frequently performed in the final weeks of pregnancy to assess fetal health. However, during the NST, the mother lies motionless in a supine position for approximately 20 minutes, during which time she attempts to obtain sufficient data on the baby's heart rate and movements, which can cause stress and anxiety in some women. A prolonged duration or a non-reactive test result can be a cause for concern. Therefore, simple and effective methods are needed to reduce maternal stress during the NST. Humorous and cute content, especially animal videos, are known to evoke positive emotions and provide psychological relief in viewers. The purpose of this study was to evaluate the effect of watching a cat video during the NST procedure on stress parameters and fetal physiological parameters in primiparous pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are primiparous,
* Able to communicate in Turkish,
* In their 34th-40th weeks of pregnancy,
* Have no problems that would prevent them from viewing visual or auditory materials,
* Have the cognitive ability to understand interactive video content,
* Have not engaged in physical exercise for at least 2 hours prior to fetal heart rate monitoring will be included in the study.

Exclusion Criteria:

* Pregnant women with multiple pregnancies,
* Uterine contractions detected during NST,
* Diagnosed with a high-risk pregnancy (preeclampsia, gestational diabetes, placenta previa, etc.),
* A phobia of cats (ailurophobia),
* Pregnant women who became pregnant using assisted reproductive technologies (ART),
* Have a history of a diagnosed endocrinological (e.g., hypothyroidism, hyperthyroidism, Cushing's syndrome) or psychiatric (e.g., anxiety disorder, depression) disease will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
The effect of watching cat videos on stress parameters in pregnant women | This procedure will be performed during the NST for pregnant women experiencing their first pregnancy and who are between weeks 34 and 40 of gestation.
  Participants randomly assigned to the intervention group will be taken to a designated room determined by the researcher before the NST for their initial measurements. The "Pregnant Women Demographic Information Form" and the "State-Trait Anxiety Inventory (STAI Form TX-1)" will be administered. Blood pressure, heart rate, oxygen saturation, cortisol, and ACTH levels will be measured. All physiological measurements except ACTH and cortisol will be performed at three time points: before the NST (2 minutes before start), in the middle of the NST (approximately 10 minutes), and after the NST (2 minutes after completion). The "State-Trait Anxiety Inventory (STAI Form TX-1)" will also be administered after the NST. Following the NST, satisfaction levels will also be assessed using the Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
The effect of watching cat videos on physiological parameters of the fetus | This procedure will be performed during the NST for pregnant women experiencing their first pregnancy and who are between weeks 34 and 40 of gestation.
  Participants randomly assigned to the intervention group will be taken to a designated room determined by the researcher before the NST for their initial measurements. The fetal heart rate and reactivity will be assessed using the NST device. To determine fetal well-being, the Non-Stress Test-Baseline, Non-Stress Test-Variability, Non-Stress Test-Acceleration, and Non-Stress Test-Deceleration numbers will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No